CLINICAL TRIAL: NCT01324323
Title: A Phase I Open-label, 2-period Study to Evaluate the Influence of Multiple Oral Doses of Rifampin on the Single Dose Pharmacokinetics of Romidepsin in Subjects With Advanced Cancer
Brief Title: Influence of Rifampin on the Pharmacokinetics of Romidepsin in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ROMI-ADVM-002; 2010-022149-75 (EudraCT Number)
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Hematologic Malignancy; Malignant Lymphoma
Keywords: ROMI-001; romi; Romidepsin; Istodax; advanced malignancy; PK; pharmacokinetics
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma | interventions — romidepsin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romidepsin and rifampin (Experimental): Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8.
  Rifampin 600 mg oral once daily on Days 4-8
  Interventions: Drug: Romidepsin; Drug: Rifampin

INTERVENTIONS:
Drug: Romidepsin — 14 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8.
  Other Names: Istodax®, Romi, ROMI
Drug: Rifampin — 600 mg oral once daily on Days 4-8

SUMMARY:
The purpose of this study is to evaluate the effect and safety of multiple doses of rifampin on the pharmacokinetics of romidepsin after a single intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older at the time of signing the informed consent document.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Must have diagnosis of advanced malignancy and must have failed other available therapies considered standard of care for their disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Negative urine or serum pregnancy test on females of childbearing potential; and
7. All females of childbearing potential must use an effective barrier method of contraception (either an intrauterine contraceptive device [IUCD] or double barrier method using condoms or a diaphragm plus spermicide) during the treatment period and for at least 1 month thereafter. Male subjects should use a barrier method of contraception during the treatment period and for at least 3 months thereafter. Female subjects should avoid the use of estrogen-containing contraceptives, since romidepsin may reduce the effectiveness of estrogen-containing contraceptives. An in vitro binding assay determined that romidepsin competes with β-estradiol for binding to estrogen receptors.

Exclusion Criteria:

1. Any significant medical condition or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subjects with significant gastrointestinal disease that may impair drug absorption, such as subjects with a history of Cohn's disease, colectomy, gastrectomy, celiac disease, or other diseases with known malabsorption.
4. Serum potassium < 3.8 mmol/L or serum magnesium < 0.85 mmol/L (magnesium converts to 2.1 mg/dl or 1.7 mEq/L) (electrolyte abnormalities can be corrected with supplementation to meet inclusion criteria).
5. Concomitant use of drugs that may cause a significant prolongation of the corrected measurement of the time between the start of the cardiac Q wave and the end of the T wave (QTc).
6. Concomitant use of Cytochrome P 450 3A4 (CYP3A4) strong inhibitors within 1 week of trial medications.
7. Concomitant use of CYP3A4 strong inducers within 2 weeks of trial medications.
8. Concomitant use of therapeutic warfarin due to a potential drug interaction. Use of a low dose of warfarin or another anticoagulant to maintain patency of venous access port and cannulas is permitted.
9. Clinically significant active infection.
10. Known infection with Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C.
11. Inadequate bone marrow or other organ function as evidenced by:

    * Hemoglobin < 9 g/dL (transfusions and/or erythropoietin are permitted);
    * Absolute neutrophil count (ANC) ≤ 1.0 * 10^9 cells/L [subjects with neutropenia (ANC 1-1.5) as a function of their disease may be supported with granulocyte-colony stimulating factor (G-CSF)];
    * Platelet count < 100 * 10^9 cells/L or platelet count < 75 * 10^9 cells/L if bone marrow disease involvement is documented;
    * Total bilirubin > 1.5 * upper limit of normal (ULN) or > 2.0 * ULN in the presence of demonstrable liver metastases;
    * Serum aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) > 1.5 * ULN or > 2.0 * ULN in the presence of demonstrable liver metastases; or
    * Serum creatinine > 2.0 * ULN;
12. Prior chemotherapy treatment within 3 weeks prior to the first day of romidepsin treatment (6 weeks for nitrosoureas) or prior treatment with an investigational agent within 4 weeks prior to the first day of romidepsin treatment.
13. Prior radiotherapy within 4 weeks prior to the first day of treatment. Subjects who have not fully recovered or whose acute toxicity related to prior radiotherapy has not returned to baseline are ineligible.
14. Major surgery within 2 weeks of study entry (day 1).
15. Concomitant use of any other anti-cancer therapy.
16. Concomitant use of any investigational agent.
17. Prior exposure to romidepsin (other histone deacetylase [HDAC] inhibitors are allowed).
18. Any known cardiac abnormalities, such as:

    * Congenital long measure of the time between the start of the Q wave and the end of the T wave (QT) syndrome;
    * Mean QTc formula (QTcF) interval > 450 msec;
    * A myocardial infarction within 12 months of study entry;
    * A history of coronary artery disease (CAD), e.g., angina Canadian Class II-IV. A stress imaging study should be performed for any subject whose cardiac status is uncertain. If abnormal, an angiography should be completed to define whether or not CAD is present.
    * An electrocardiogram (ECG) recorded at screening showing evidence of cardiac ischemia (ST depression of ≥ 2 mm, measured from isoelectric line to ST segment). A stress imaging study should be performed for any subject whose cardiac status is uncertain. If abnormal, an angiography should be completed to define whether or not CAD is present.
    * Congestive Heart Failure (CHF) that meets the New York Heart Association (NYHA) Class II to IV definitions (see Appendix F) and/or ejection fraction < 40% by multi gated acquisition (MUGA) scan or < 50% by echocardiogram and/or magnetic resonance imaging (MRI);
    * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), torsades de pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
    * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes (if in doubt, see ejection fraction criteria above);
    * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥ 160/95; or
    * Any cardiac arrhythmia requiring anti-arrhythmic medication.
19. Subjects who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2012-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Takeshita, MD, Study Director — Celgene Corporation
Locations (3):
- United States (2):
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Canon Research Institute, Nashville, Tennessee
- Sarah Cannon Research UK, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 study centers (2 in the United States and 1 in the United Kingdom). The first subject was enrolled in April 2011 and the last subject completed the study in Feb 2012.
Period: Overall Study
Arm/Group | Romidepsin and Rifampin
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Romidepsin and Rifampin
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 13
  Black or African American | 1
  Other | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5
  United States | 9
Height [Mean (Standard Deviation); unit: Centimeters] | 167.6 (9.54)
Weight [Mean (Standard Deviation); unit: kilograms] | 78.2 (18.85)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: Metered Squares m^2] | 1.9 (0.22)
Eastern Cooperative Oncology Group Performance Status (ECOG) [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living activities of the patient and determine appropriate treatment and prognosis.
  0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully active | 7
    1 = Restricted in physical strenuous activity | 7
    2 = Ambulaotry but unable to work | 0
    3 = Limited Self-Care | 0
    4 = Completely Disabled | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time-curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-t)of Romidepsin
Description: AUC0-t: area under the plasma concentration time-curve from Time 0 to the time of the last quantifiable concentration (Ct), calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: Days 1 and 8; at 0 (pre-dose), 1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion.
Population: The PK population included all participants who received at least 1 dose of study drug and had evaluable PK profiles. The primary reason for study discontinuation for the 1 participant was due to withdrawal of consent.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Romidepsin Day 1: Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8.
- Romidepsin and Rifampin Day 8: Romidepsin 14mg/m^2 intravenous infused over 4 hours on Day 8. Rifampin 600mg oral once daily on Days 4-8.
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
ng*hr/mL | 2225.1 (71.4) | 3966.3 (76.5)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Rifampin Day 8; Test type: Superiority or Other; ANOVA; Ratio of the Geometric Mean (%) = 179.3, 90% CI 2-sided [160.3 to 200.7] — Ratio ("Romidepsin + rifampin"/"Romidepsin") and 90% CI of the ratio of geometric means are from an ANOVA model with treatment as fixed effect and subject as random effect on the natural log transformed PK values

2. Primary Outcome: Area Under the Plasma Concentration Time-curve From Time 0 to 24-hour (AUC0-24) for Romidepsin
Description: Individual and mean romidepsin plasma concentrations by treatment and scheduled time data were collected. AUC0-24: area under the plasma concentration time-curve from Time 0 to 24 hours, calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: Day 1 and Day 8; at 0 (predose), 1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Romidepsin Day 1: Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Day 1.
  Rifampin 600 mg oral once daily on Days 4-8
- Romidepsin and Rifampin Day 8: Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Day 8. Rifampin 600 mg oral once daily on Days 4-8
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
ng*hr/mL | 2204.2 (72.0) | 3903.9 (78.0)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Rifampin Day 8; Test type: Superiority or Other; ANOVA; Ratio of the Geometric Mean = 178.3, 90% CI 2-sided [159.4 to 199.4] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Plasma Concentration Time-curve From Time Zero Extrapolated to Infinity (AUC0-∞).
Description: AUC0-∞: area under the plasma concentration time-curve from Time 0 extrapolated to infinity, calculated as [AUCt + Ct/λz]. λz is the apparent terminal rate constant. No AUC extrapolation was performed with unreliable λz. If the percentage of AUC extrapolated is ≥ 25%, AUC0-∞ will not be reported.
Time Frame: Days 1 and 8; at 0 (predose), 1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion.
Population: The primary objective was to assess the influence of multiple doses of rifampin on the PK of romidepsin. The PK population included all participants who received at least 1 dose of study drug and had evaluable PK profiles. The primary reason for study discontinuation for the 1 participant was due to withdrawal of consent.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Romidepsin Day 1: Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Day 1
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
ng*hr/mL | 2229.8 (71.3) | 3980.7 (76.1)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Rifampin Day 8; Test type: Superiority or Other; ANOVA; Ratio of the Geometric Mean = 179.6, 90% CI 2-sided [160.5 to 201.0] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)of Romidepsin
Description: Maximum observed plasma concentration (Cmax)was obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Romidepsin and Rifampin Day 8: Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Day 8. Rifampin 600mg oral once daily on Days 4-8
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
ng/mL | 571.2 (81.0) | 900.1 (104.9)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Rifampin Day 8; Test type: Superiority or Other; ANOVA; Ratio of the Geometric Mean = 159.1, 90% CI 2-sided [135.8 to 186.5] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax)
Description: Time to maximum observed plasma concentration (Tmax) was obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
hours | 3.0 (51.5) [1.00 to 5.00] | 3.00 (50.7) [1.00 to 4.27]
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Rifampin Day 8; Note: The median, median difference ("romidepsin + rifampin" minus "romidepsin") and 90% CI of the median difference are from Hodges-Lehmann Estimate. The P-value is from Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.7910, Wilcoxon signed-rank; Median Difference (Final Values) = -0.15, 90% CI 2-sided [-1.0 to 1.01]

6. Primary Outcome: Estimate of the Terminal Elimination Half-life in Plasma (t1/2)
Description: The terminal elimination half-life (t1/2) in plasma, was calculated as [(ln 2)/λz]. This was only calculated when a reliable estimate for λz could be obtained.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
hours | 9.666 (27.9) | 8.341 (24.0)

7. Primary Outcome: Clearance (CL): Apparent Total Plasma Clearance.
Description: The apparent total plasma clearance (CL) was calculated as [Dose/AUC0-∞] for Romidepsin alone and co-administered with rifampin plasma concentrations.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
L/hr | 11.59 (78.1) | 6.45 (82.2)

8. Primary Outcome: Apparent Total Volume of Distribution (Vz).
Description: Apparent total volume of distribution (Vz) was calculated as [(CL)/λz] for Romidepsin and co-administered with Rifampin.
Time Frame: as for outcome 3
Population: The PK population was to consist of all participants who received at least 1 dose of study drug and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Romidepsin Day 1 | Romidepsin and Rifampin Day 8
Number analyzed (Participants) | 14 | 13
Liters | 161.48 (78.6) | 77.6 (93.8)

9. Secondary Outcome: Summary of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: AEs were considered related if assessed by the Investigator as possibly, probably or definitely related to study drug. Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Day 1 up to Day 36 (28 days after the last treatment)
Population: The safety population included all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Romidepsin Plus Rifampin: Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Days 1 and 8. Rifampin 600 mg oral once daily on Days 4-8
Arm/Group | Romidepsin Plus Rifampin
Number analyzed (Participants) | 14
participants
  = > 1 TEAE | 13
  = > 1 TEAE related to any study drug | 13
  = > 1 TEAE related to Romidepsin | 13
  = > 1 TEAE related to Rifampin | 2
  = > 1 Serious TEAE | 2
  = > 1 Serious TEAE related to any drug | 1
  = > 1 Serious TEAE related to Romidepsin | 1
  = > 1 Serious TEAE related to Rifampin | 1
  = > 1 TEAE leading to discontinuation | 0
  = > 1 TEAE related discontinuation to any drug | 0
  = > 1 Romidepsin related TEAE discontinuation | 0
  = > 1 Rifampin related TEAE discontinuation | 0
  Participants who died | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 36 (28 days after last treatment)
Groups:
- Romidepsin Plus Rifampin: Romidepsin 14 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8 and Rifampin 600 mg oral once daily on Days 4-8.
Arm/Group | Romidepsin Plus Rifampin
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin Plus Rifampin (N=14)
Anaemia (Blood and lymphatic system disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Melaena (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin Plus Rifampin (N=14)
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Asthenia (General disorders) | 1
Malaise (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 3
Decreased Appetite (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation